CLINICAL TRIAL: NCT05896150
Title: Intercostal Cryoanalgesia for Management of Acute Postoperative Pain Following Video-assisted Thoracoscopic Lung Cancer Resection
Brief Title: Intercostal Cryoanalgesia for Acute Pain After VATS Lung Resection
Acronym: CRYO-VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-11561
Record Dates: First submitted 2023-05-19; First posted 2023-06-09 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Thoracic Surgery; Video-Assisted; Cryotherapy Effect; Paravertebral Block

STUDY DESIGN:
Intervention Model Description: Intervention : intercostal cryoanalgesia + single-injection paravertebral block Control group : single-injection paravertebral block
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostal cryoanalgesia AND single-injection paravertebral block (Experimental): * Videothoracoscopic-guided single-injection paravertebral block at T5 with 0.4 mL/kg of Bupivacaine 0.5% with adrenalin 5 mcg/mL (maximum 40 mL) at the beginning of surgery
  * Cryoanalgesia 5 cm lateral to the neuraxial, on the inferior costal border, CO2 at (-)50C to (-)70C for 2 minutes, repeated on 7 costal levels (T3-T9), after the lung resection and before chest closure.
  Interventions: Procedure: Cryoanalgesia AND single-injection paravertebral block
- Single-injection paravertebral block (Active Comparator): -Videothoracoscopic-guided single-injection paravertebral block at T5 with 0.4 mL/kg of Bupivacaine 0.5% with adrenalin 5 mcg/mL (maximum 40 mL) at the beginning of surgery
  Interventions: Procedure: Single-injection paravertebral block

INTERVENTIONS:
Procedure: Cryoanalgesia AND single-injection paravertebral block — CO2 Cryoanalgesia AND paravertebral block with Bupivacaine 0.5%
  Arms: Intercostal cryoanalgesia AND single-injection paravertebral block
Procedure: Single-injection paravertebral block — Paravertebral block with Bupivacaine 0.5%
  Arms: Single-injection paravertebral block

SUMMARY:
Intercostal cryoanalgesia is a technique that allows extensive and prolonged analgesia of the hemithorax. The aim of this study is to demonstrate the efficacy of intercostal cryoanalgesia as an adjunct to a single-injection paravertebral block for the management of acute thoracic pain after VATS lung resection surgery.

DETAILED DESCRIPTION:
VATS lung resection is associated with a high incidence of moderate to severe acute thoracic pain. In the postoperative period, optimal analgesia may facilitate recovery, lead to higher patient satisfaction, and lower postoperative complications.

Regional analgesia techniques are usually recommended for VATS, and the paravertebral block is often used. However, the duration of the paravertebral block is short (6 to 24 hours), and prolongation of the effect requires the placement of a paravertebral catheter and local anesthetic infusion into the paravertebral space. At our institution, patients with VATS lung resections are often discharged home 24-48 hours after surgery.

Intercostal cryoanalgesia has an onset of about 12 hours, which coincides with the weaning of the single-injection paravertebral block. Analgesia is usually prolonged over several weeks, does not require catheter placement, and is not associated with hemodynamic side effects. These characteristics may allow rapid recovery and safe home discharge after VATS lung resection.

The aim of this study is to demonstrate the efficacy of intercostal cryoanalgesia as an adjunct to a single-injection paravertebral block for the management of acute thoracic pain after VATS lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective anatomical pulmonary resection (anatomical segmentectomy, lobectomy or bilobectomy) by VATS for lung cancer
* American Society of Anesthesiologists (ASA) score 1-3

Exclusion Criteria:

* Contraindication to the paravertebral block (coagulopathy, discontinuous paravertebral space, impossible thoracoscopic visualization of the paravertebral space)
* Contraindication to intercostal cryoanalgesia (cold urticaria, cryoglobulinemia)
* Epidural analgesia preferred (high risk of thoracotomy, marginal lung function)
* Surgical criteria (conversion to thoracotomy, non anatomical wedge resection)
* Known allergy to acetaminophen, celecoxib, sulfa or both hydromorphone and morphine
* Preoperative thoracic or shoulder pain on the operated side
* History of thoracic surgery on the operated site
* Regular use of opioids or medication with effects against neuropathic pain (tricyclics, gabapentinoids, duloxetine, venlafaxine)
* Inability to understand pain scales or to communicate clearly despite adequate teaching
* Contraindication to non-steroidal anti-inflammatory drugs (renal filtration rate < 60 mL/min, active gastric ulcer)
* Pregnancy
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Acute thoracic pain during cough | 24 hours
  Numerical Rating Scale (NRS) score : scale 0 (no pain) to 10 (worst)

SECONDARY OUTCOMES:
Acute thoracic pain at rest | 1 hour, 6 hours, 12 hours, 18 hours, 24 hours, 48 hours and 7 days
  Numerical Rating Scale (NRS) score : scale 0 (no pain) to 10 (worst)
Acute thoracic pain during cough | 1 hour, 6 hours, 12 hours, 18 hours, 48 hours and 7 days
  Numerical Rating Scale (NRS) score : scale 0 (no pain) to 10 (worst)
Postoperative morphine-equivalents consumption | 7 days
  Using a Patient Controlled Analgesia (PCA) pump for the first 24 hours, then daily
QoR-15 score : 0 (worst) to 150 (best) | Preoperative and 48 hours postoperative
  QoR-15 is a score evaluating the quality of recovery after surgery and anesthesia
Hypoesthesia over the ipsilateral thorax | 24 hours
  Evaluation of the dermatomal levels of hypoesthesia using a Von Frey monofilament
Incidence of nausea related to opioid consumption | 7 days
  Evaluation for nausea (yes or no)
Time to hospital discharge | 30 days
  Total time between the end of surgery and prescription for hospital discharge
Evaluation of sedation related to opioid consumption | 7 days
  Using the Ramsay score (1 to 6)
Incidence of vomiting related to opioid consumption | 7 days
  Evaluation for vomiting (yes or no)
Incidence of pruritus related to opioid consumption | 7 days
  Evaluation for pruritus (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Moore, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal
Locations (1):
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No